CLINICAL TRIAL: NCT00882492
Title: Identifying a Novel Mechanism for Perioperative Hyperglycemia Identifying a Novel Mechanism for Perioperative Hyperglycemia in Cardiac Surgery: A Role for Incretins
Brief Title: GLP 1 for Intraoperative Glycemic Control
Acronym: GLP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP 1 01
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Hyperglycemia; Hypoglycemia
Keywords: Cardiac; Surgery; Glycemia
MeSH Terms: conditions — Hyperglycemia; Hypoglycemia | interventions — Glucagon-Like Peptide 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): This active arm is a continuous infusion of GLP-1 during cardiac surgery
  Interventions: Biological: GLP 1
- 2 (Placebo Comparator): This is a continuous infusion of normal saline solution infusion as placebo at (1.5 pmol/kg/min)
  Interventions: Biological: normal saline solution placebo

INTERVENTIONS:
Biological: GLP 1 — This a continuous intravenous infusion of GLP-1 (7-36) amide infusion (1.5 pmol/kg/min)
  Arms: 1
Biological: normal saline solution placebo — This is a continuous intravenous infusion of normal saline solution as placebo (1.5 pmol/kg/min) during cardiac surgery
  Arms: 2

SUMMARY:
This is a medical research study designed to see if an infusion of a naturally occurring hormone, GLP-1, works when used to decrease blood sugar during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. male or female age (18-80 years),
2. ability to provide informed consent,
3. elective CABG with or without single or multivalve repair or replacement, and/ or
4. single or multivalve repair or replacement requiring CPB and sternotomy (to include subjects who are undergoing first time or redo cardiac surgery).

Exclusion Criteria:

1. concomitant surgery (e.g. carotid endarterectomy),
2. emergent surgery,
3. current steroid use,
4. insulin dependent diabetes mellitus (IDDM),
5. cardiac surgery without the use of cardiopulmonary bypass (e.g. off-pump CABG),
6. current use of positive intravenous inotropic agents,
7. serious intercurrent illness (endocarditis, sepsis, active malignancy requiring treatment) or active infection,
8. known substance abuse,
9. receipt of an investigational drug or device within 30 days prior to surgery,
10. known allergy to any of the following: GLP-1, fentanyl, midazolam, isoflurane, propofol, morphine, heparin or protamine,
11. Sulfonylurea medication administration on morning of surgery (such as, tolbutamide, tolazamide (Tolinase), chlorpropamide (Diabinese). glipizide (Glucotrol, Glucotrol XL), glyburide (Micronase, Glynase PresTabs, and DiaBeta), glimepiride (Amaryl),
12. Major end organ dysfunction defined as:

    1. Cardiac: Left ventricular ejection fraction (LVEF) < 30% by left ventriculography or echocardiogram (within 90 days prior to randomization), current use of positive intravenous inotropic agents, preoperative use of intra-aortic balloon pump (IABP), left ventricular assist device (LVAD), or extracorporeal membrane oxygenation (ECMO);
    2. Renal: preoperative serum Creatinine > 2.0 mg/dL;
    3. Hepatic: aspartate aminotransferase (AST) or alanine transferase (ALT) > 2.5 x upper limit normal;
    4. Hematologic: preoperative hematocrit (HCT) < 30%, platelet count < 100,000/mm3, history of (or family history of) bleeding or clotting disorder;
13. Patients with a history of or risk factors for acute pancreatitis (i.e. ethanol abuse, gall stones) will be excluded from this study,
14. Pregnant or breastfeeding females, or
15. any other condition that, in the opinion of the investigator, may compromise the safety of the subject or would preclude the subject from successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome variables are plasma GLP-1 levels and plasma Glucose levels. | During surgery and 24 hours after

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States